CLINICAL TRIAL: NCT04114474
Title: Pre-operative Focused Transthoracic Echocardiography for Prediction of Post-operative Cardiac Complications
Status: Completed | Type: Observational
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Alaa Ali M. Elzohry, Lecturer of Anesthesia, ICU and Pain Relief, South Egypt Cancer Institute, Assiut University., South Egypt Cancer Institute
Other Study IDs: transthoracic echocardiograpy
Record Dates: First submitted 2019-09-27; First posted 2019-10-03 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Diastolic Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: TRANSTHORACIC ECHOCARDIOGRAPY — TTE (Vivid I echocardiography machine General Electric Healthcare, Milwaukee, WI, USA) with a 3S-RS (1.5-3.6 MHz) transthoracic probe). was done by professional anesthesiologist following the :Hemodynamic Echocardiography Assessment in Real Time ( HEART) protocol. According to the clinical findings of TTE patients may be either free or have one or more of the following haemodynamic states normal, empty, vasodilated ,left ventricular systolic or diastolic failure, left ventricular systolic and diastolic failure, and right ventricular failure, valve stenosis or regurgitation of at least moderate severity

SUMMARY:
The extent focused transthoracic echocardiography when done pre-operatively to patients admitted for elective surgery and suspected to be at risk of cardiac disease specially the geriatric population can affect perioperative anesthetic management of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 60 years of age ASAI and ASA II were included

Exclusion Criteria:

* history of cardiac disease, history of previous postoperative cardiac complications and symptoms or signs of cardiac diseases.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligibility for participating in the study was assessed before assignment by the attending physician in the anesthesia clinic . Patients above 60 years of age ASAI and ASA II were included in the study unless history of cardiac disease, history of previous postoperative cardiac complications and symptoms or signs of cardiac diseases were found as theses patients were excluded from the study.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Lt. Ventricular EDV | Change from Baseline pre operative LVEDV to first day postoperative
  Transthoracic echocardiography (TEE) LVEDV

CONTACTS AND LOCATIONS:
Overall Officials: ALAA A EALZOHRY, MD, Principal Investigator — Lecturer of Anesthesia, ICU and Pain Relief, South Egypt Cancer Institute.
Locations (1):
- South Egypt Cancer Institute, Assiut University, Arab Republic of Egypt, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT04114474/Prot_SAP_000.pdf